CLINICAL TRIAL: NCT07194720
Title: Effects of the Cornelian Cherry (Cornus Mas L.) Lyophilisate Supplementation on the Selected Physiological Parameters in Amateur Long-Distance Runners
Brief Title: Effects of the Cornelian Cherry Supplementation on the Selected Physiological Parameters in Marathon Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Collaborators: Wrocław University of Environmental and Life Sciences (Unknown)
Responsible Party: Principal Investigator, Rafał Seredyński, Principal Investigator, Wroclaw Medical University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: DEREN.23.25
Record Dates: First submitted 2025-09-18; First posted 2025-09-26 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Cornus mas L.; systemic vascular resistance; peripheral chemoreflex; endurance training; nitric oxide; endothelium; autonomic nervous system; blood pressure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cornus mas lyophilisate (Experimental)
  Interventions: Dietary Supplement: Cornus mas lyophilisate
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cornus mas lyophilisate — Participants receiving a Cornus mas (Cornelian cherry) lyophilisate for 4 weeks.
  Arms: Cornus mas lyophilisate
Dietary Supplement: Placebo — Participants receiving a starch- and sugar-based placebo for 4 weeks.
  Arms: placebo

SUMMARY:
Growing body of evidence indicates favorable effects of Cornus mas (Cornelian cherry) supplements on cardiometabolic risk, including the improvement of HDL and glycemic indices, in line with vascular benefits. Experimental data feature bioactives from Cornelian cherry as potential modulators of vascular function and blood pressure, plausibly via endothelial nitric oxide-related pathways, with possible downstream effects on autonomic reflex control; nevertheless, such links in humans remain poorly explored to date, especially in terms of endurance training and hypoxia tolerance.

In this cross-over, placebo-controlled study, a group of healthy amateur long-distance runners underwent two stages of a four-week dietary intervention (separated by four weeks of washout period), receiving Cornelian cherry lyophilisate or placebo. Each supplementation stage was accompanied by the comprehensive evaluation of the cardio-respiratory parameters and endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* age above 45 years

Exclusion Criteria:

* chronic disease of the nervous, cardiovascular or respiratory system
* disease of the digestive system, including history of the intestinal surgery, inflammatory bowel disease, celiac disease, lactose intolerance and other malabsorption disorders
* blood pressure-lowering treatment within the past year
* tobacco smoking within the past year
* antibiotic/probiotic treatment and laxative/prokinetic usage in three months preceding the anticipated enrollment

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
Systemic vascular resistance | From the beginning to the end of a supplementation period at 4 weeks.
  Resting systemic vascular resistance, evaluated non-invasively with a finger cuff-based device.
Office blood pressure values (mean, systolic, diastolic) | From the beginning to the end of a supplementation period at 4 weeks.
  Resting arterial blood pressure values (mean, systolic, diastolic), measured continuously with a non-invasive, finger cuff-based device.

SECONDARY OUTCOMES:
Peripheral chemoreflex sensitivity | From the beginning to the end of a supplementation period at 4 weeks.
  Peripheral chemoreflex sensitivity, measured with the transient hypoxia test.
eNOS expression | From the beginning to the end of a supplementation period at 4 weeks.
  Endothelial nitric oxide synthase expression, evaluated in the peripheral blood samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Wroclaw Medical University, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
This is a small trial which includes solely healthy volunteers. Therefore, data will not be shared at this instance.